CLINICAL TRIAL: NCT03760172
Title: Immunomediated Non-alcoholic SteaTohepatitis; Prevalence and Characterization. INSTInCT Study
Acronym: INSTInCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Hospital Universitario La Fe (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, MARIA CINTA ALMENARA MIRAMON, Dr. Javier Crespo Garcia, Instituto de Investigación Marqués de Valdecilla
Other Study IDs: PI18/01304
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Main Hypothesis is That in the NASH Associated to IMIDs, to Different Phenotypes co Exist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prevalence of NAFLD in patients with IMID: To analyze the global prevalence of NAFLD in patients with an immune-mediated inflammatory disease IMID
- Prevalence of High-risk NASH in patients with IMID: To evaluate the prevalence of high-risk NASH (NASH with advanced fibrosis) in patients with IMID through clinical, radiological and histological evaluation
- Immunophenptypic characterization: To investigate the existence of common and differential immunophenotypes between the subjects with NASH with and without IMID, and patients with IMID without liver involment
- Genetic and Molecular characterization: Liver molecular characterization of NASH associated to IMID

SUMMARY:
NAFLD is a common comordidity in patients with IMID, including inflammatory bowel disease and psoriasis.

Nevertheless, the prevalence of NAFLD and NASH in the IMID population is not clear, and the risk factors are not completely understood. Interestingly, NASH and most of IMIDs share main molecular and immunological mechanisms of disease, as the inflammatory pathways depending on TNFa or imbalance in T cell subtypes like Th17/Treg. This common pathogenesis may explain, at least in a subset of patients, the development of NASH in the absence of classic metabolic risk factor.

Thus, our main hypothesis is that in the NASH assciated to IMIDs two different phenotypes co-exist.

First, a predominantly inflammatory phenotype, and not associated to the metabolic syndrome ande second, a predominantly metabolic phenptype, strongly associated to he metabolic syndrome.

In this way, we believe that in a particular subset of NAFLD patients, NASH could be considered as an IMID, as most of the definiting features of IMIDs are present. To demonstrate our hypothesis, we consider a two-stage study. First, we will determine the NAFLD and NASH prevalence in a cohort of well-characterized IMID patients and controls. Second, we will adress the molecular and immunophenotype characterization in liver biopsies of NASH patients with and without the co-existence of IMIDs.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD with biopsy proven disease above 18 years
* IMID patients above 18 years
* All participants must give informed written consent

Exclusion Criteria:

* Patients who had any clinical evidence of malignancy
* Other secondary cause of chronic liver disease. Alternative causes of liver disease included excessive alcohol intake (higher than 20 g/day in women and 30 g/day in men), viral hepatitis, chronic alcohol consumption, autoimmune hepatitis, Wilson´s disease, alpha-1-antitripsine deficiency, inborn errors of metabolism or drug induced liver injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all population
Sampling Method: Non-Probability Sample
Enrollment: 7300 (Estimated)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD in patients with IMID | January 2019 - December 2020
  Prevalence of NAFLD in patients with IMID

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marques de Valdecilla, Santander, Cantabria, Spain